CLINICAL TRIAL: NCT05831826
Title: Multicenter Clinical and Basic Research on the Prevention and Treatment of 2019-nCoV by Integrated Traditional Chinese and Western Medicine
Brief Title: Effectiveness and Safety of the Inactivated COVID-19 Vaccine in Thousands of Patients With Autoimmune Diseases in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Chengping Wen, Professor, Zhejiang Chinese Medical University
Other Study IDs: ZhejiangCMU 2020-KL-0601-1
Record Dates: First submitted 2023-04-25; First posted 2023-04-26 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: COVID-19 Vaccines; Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples and urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy controls: Healthy controls are ≥18 years old, no previous history of SARS-CoV-2 infection, and no previous history of autoimmune diseases. All the HC group were injected with 2 or 3 doses of inactivated SARS-CoV-2 vaccines.
  Interventions: Biological: the inactivated COVID-19 vaccines
- the vaccinated patients with ADs: The vaccinated patients with ADs are ≥18 years old, no previous history of SARS-CoV-2 infection, and diagnosed with autoimmune diseases. All the group were injected with the inactivated SARS-CoV-2 vaccines.
  Interventions: Biological: the inactivated COVID-19 vaccines
- the unvaccinated patients with ADs: The vaccinated patients with ADs are ≥18 years old, no previous history of SARS-CoV-2 infection, and diagnosed with autoimmune diseases. All the group were not injected with the inactivated SARS-CoV-2 vaccines.

INTERVENTIONS:
Biological: the inactivated COVID-19 vaccines — receive the doses of inactivated COVID-19 vaccines
  Groups: healthy controls; the vaccinated patients with ADs

SUMMARY:
According to the comprehensive evaluation, the completion of vaccination and the prevention and treatment strategy of integrated traditional Chinese and western medicine have obvious advantages in improving the symptoms of infection in patients with autoimmune diseases, shortening the course of disease and controlling disease activity, and can play a positive role in the whole process of epidemic prevention and treatment. Now the investigators plan to conduct multi-center clinical and basic research to observe the preventive effect and safety of the vaccine on COVID-19, as well as the preventive effect of the combination of traditional Chinese medicine, in order to obtain high-quality evidence-based evidence and provide scientific basis for the clinical value of the drug.

DETAILED DESCRIPTION:
Autoimmune diseases are disorders of the body's immune function, involving multiple organs and tissues of the whole body, and characterized by a variety of specific or non-specific autoantibodies and inflammatory factors overexpression. However, during the global COVID-19 pandemic, patients with autoimmune diseases, especially those receiving immunosuppressive therapy, face a high burden of novel coronavirus pneumonia (COVID-19) and are at higher risk for severe infection and disease progression. At present, patients with autoimmune diseases should give priority to the prevention and treatment strategy of COVID-19, among which the vaccination of novel coronavirus vaccine is the most important means to actively build herd immunity and control the epidemic of novel coronavirus pneumonia, and the combination of traditional Chinese and western medicine is an essential and effective way to prevent and treat COVID-19 infection. According to the comprehensive evaluation, the completion of vaccination and the prevention and treatment strategy of integrated traditional Chinese and western medicine have obvious advantages in improving the symptoms of infection in patients with autoimmune diseases, shortening the course of disease and controlling disease activity, and can play a positive role in the whole process of epidemic prevention and treatment. Now the investigators plan to conduct multi-center clinical and basic research to observe the preventive effect and safety of the vaccine on COVID-19, as well as the preventive effect of the combination of traditional Chinese medicine, in order to obtain high-quality evidence-based evidence and provide scientific basis for the clinical value of the drug.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* The ADs group were diagnosed with autoimmune diseases according to the following inclusion criteria: rheumatoid arthritis (RA) / American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2010 classification criteria; ankylosing spondylitis (AS) / the 1984 modified New York criteria; systemic lupus erythematosus (SLE) / 2019 EULAR/ACR classification criteria; Sjögren's Syndrome (SS) / 2016 ACR/EULAR Classification Criteria; systemic vasculitis / Chapel Hill Consensus Conference definitions; idiopathic inflammatory myositis (IIM) / 2017 EULAR/ACR classification criteria; psoriatic arthritis (PsA) / 2006 Classification Criteria for PsA; systemic sclerosis (SSc) / 2013 ACR/EULAR collaborative initiative; polymyalgia rheumatica (PMR) / 2012 provisional classification criteria.
* The HC group were volunteers who did not have history of autoimmune diseases and did not receive immunosuppressive therapy.

Exclusion Criteria:

* history of COVID-19 infection
* history of vaccination allergy
* history of mental disabilities
* pregnancy
* unwillingness to sign informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ADs (≥18 years old) were recruited into the study according to the following inclusion criteria: rheumatoid arthritis (RA) / American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2010 classification criteria; ankylosing spondylitis (AS) / the 1984 modified New York criteria; systemic lupus erythematosus (SLE) / 2019 EULAR/ACR classification criteria; Sjögren's Syndrome (SS) / 2016 ACR/EULAR Classification Criteria; systemic vasculitis. Patients were instructed to continue taking all drugs during the vaccination period, except for biotherapy that was delayed after the vaccination by physician's suggestion. The HC were healthy volunteers who did not receive immunosuppressive therapy.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of local and systemic adverse events | 3 years
  One of the primary end point was the safety of the inactivated COVID-19 vaccine in adult patients with ADs compared with controls.
Concentration of anti-SARS-CoV-2 spike protein | 3 years
  One of the primary end point was the immunogenicity of the inactivated COVID-19 vaccine in adult patients with ADs compared with controls.
Infection rate of COVID-19 | 3 years
  One of the primary end point was the efficacy of the inactivated COVID-19 vaccine in adult patients with ADs.

CONTACTS AND LOCATIONS:
Overall Officials: Wumeng Jin, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- The Affiliated Hospital of Zhejiang Chinese Medicine University, Hangzhou, Zhejiang, China